CLINICAL TRIAL: NCT01267708
Title: Platelet Function in Patients Undergoing PCI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Ariel Roguin, Rambam
Other Study IDs: 431-10 CTIL; 431-10.2010
Record Dates: First submitted 2010-12-27; First posted 2010-12-28 (Estimated); Last update posted 2010-12-28 (Estimated); Status verified 2010-11

CONDITIONS: All PCI Patients

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group: All those tested

SUMMARY:
The purpose of this study is to examine PLT function in PCI patients.

ELIGIBILITY:
Inclusion Criteria:

* All consented patients undergoing PCI

Exclusion Criteria:

* Unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: To examine PLT function in all patients undergoing PCI to our center
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2010-11

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Medical Center, Haifa, Israel